CLINICAL TRIAL: NCT03417219
Title: Mobile Media Intervention for Family Caregivers of Veterans With Dementia
Brief Title: Mobile Tablet Education to Advance Caregiver Health
Acronym: MTEACHing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E1710-P; 1I21RX001710 (NIH)
Record Dates: First submitted 2018-01-23; First posted 2018-01-31 (Actual); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-01

CONDITIONS: Dementia
Keywords: Caregivers; Family; Veterans; Alzheimer Disease; Memory
MeSH Terms: conditions — Dementia; Alzheimer Disease | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobile Media Education and Skill-Building Rehabilitation Int (Experimental): The investigators' ESBR-m intervention consists of four, 90-minute group (= 5 participants) sessions. These four sessions are supplemented with a booster session one month following the last intervention session.
  Interventions: Behavioral: Education and Skill Building Rehabilitation-mobile (ESBR-m)
- Usual Care (Active Comparator): Usual Care (plus supplemental educational materials). Participants randomized to the Usual Care (UC) group will receive supplemental educational materials (e.g., VA Caregiver Support Program; Veterans Crisis Line; National Institute on Aging's "Understanding Memory Loss").
  Interventions: Behavioral: Usual Care (UC)

INTERVENTIONS:
Behavioral: Education and Skill Building Rehabilitation-mobile (ESBR-m) — Participants randomized to the ESBR-m group will participate in four, 90-minute group ( 5 participants) sessions. These four sessions are supplemented with a booster session one month following the last intervention session.
  Arms: Mobile Media Education and Skill-Building Rehabilitation Int
Behavioral: Usual Care (UC) — Participants randomized to the UC group will receive supplemental educational materials (e.g., VA Caregiver Support Program; Veterans Crisis Line; National Institute on Aging's "Understanding Memory Loss").
  Arms: Usual Care

SUMMARY:
To address the high burden of caring for a Veteran with dementia, the investigators propose to study the effect of a low-cost, rehabilitative intervention for family caregivers of Veterans with dementia. The investigators' novel approach will use mobile media technology that can reach caregivers in rural areas who do not have easy access to major VA medical centers. If this rehabilitative intervention proves successful, it may represent an approach to Veteran and family-centered dementia care that can be used throughout VA with low staff, resource, and cost burdens.

DETAILED DESCRIPTION:
The proposed project studies the effects of an education and skill-building rehabilitation intervention, designed to be low-cost and clinically translatable through mobile media devices (i.e., tablets), on family caregivers of Veterans with dementia. Intervention effects will be examined longitudinally at baseline and 3 months post-intervention.

Advanced statistical techniques will be used to determine the impact of the intervention on: quality of life in caregivers of Veterans with dementia (Aim 1), perceived stress and depressive symptoms in caregivers (Aim 2), and socialization and engagement in pleasant activities in caregivers (Aim 3).

If this rehabilitative intervention proves successful, it may represent an approach to Veteran- and family-centered dementia care that can be used throughout VA with low staff, resource, and cost burdens.

ELIGIBILITY:
Inclusion Criteria:

-- Participants must:

* report distress associated with being the primary caregiver for a family member with dementia
* reporting at least 2 of the following 6 items at baseline assessment: felt overwhelmed, felt like they often needed to cry, were angry or frustrated, felt they were cut off from family or friends, reported moderate to high levels of general stress, or felt their health had declined
* provide at least 7 hours of care (supervision or direct assistance) per week over the past 3 months (other sources of caregiving for the Veteran with dementia can also be utilized; e.g., respite, home health aide, other family members)
* cohabitate with a Veteran diagnosed with dementia
* be proficient in spoken and written English
* be capable of providing informed consent

Exclusion Criteria:

-- Potential participants will be screened and excluded for:

* current or lifetime history of any psychiatric disorder with psychotic features
* prominent suicidal or homicidal ideation
* having met DSM-IV criteria for drug or alcohol abuse or dependence (except nicotine) within the past six months
* presence of alcohol intoxication (by breathalyzer) or alcohol withdrawal (by exam) during study recruitment or participation
* diagnosis of probable or possible dementia
* a Telephone Cognitive Screen score of < 20
* participation in another caregiver intervention study within the past year
* lack of access to telephone and internet services in the home
* illness that would prevent study participation
* planned transfer of care receiver to another caregiver or nursing home within 6 months
* currently living with an implantable cardioverter defibrillator or pacemaker
* known pregnancy at time of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Blake K Scanlon, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Mobile Media Education and Skill-Building Rehabilitation Int: The investigators' ESBR-m intervention consists of four, 90-minute group (<= 5 participants) sessions. These four sessions are supplemented with a booster session one month following the last intervention session.
  Education and Skill Building Rehabilitation-mobile (ESBR-m): Participants randomized to the ESBR-m group will participate in four, 90-minute group ( 5 participants) sessions. These four sessions are supplemented with a booster session one month following the last intervention session.
Period: Overall Study
Arm/Group | Mobile Media Education and Skill-Building Rehabilitation Int | Usual Care
Started | 8 | 8
Completed | 8 | 5
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Media Education and Skill-Building Rehabilitation Int | Usual Care | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (10.18) | 61.12 (7.54) | 66.06 (10.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  White | 6 | 3 | 9
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Zarit Burden Interview (ZBI) at 4 Months
Description: The Zarit Burden Interview (ZBI) is a 22-item self-report measure of caregiver burden. Several version of the ZBI have been used successfully as outcome measures in interventions for dementia caregivers. Scores for each item range from 0 (never) to 4 (nearly always) on questions such as "Do you feel embarrassed by your relative's behavior?." Total scores are calculated by summing all responses and range from 0-88. A higher score is indicative of a worse outcome.
Time Frame: Baseline, 4 month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Media Education and Skill-Building Rehabilitation Int | Usual Care
Number analyzed (Participants) | 8 | 5
score on a scale | -2.25 (7.80) | 0.80 (13.48)

2. Primary Outcome: Change From Baseline Center for Epidemiological Studies-Depression (CES-D) at 4 Months
Description: The Center for Epidemiological Studies-Depression (CES-D) is a 20-item, self-report measure of frequency of depressive symptoms over a one week period. The CES-D is frequently used to assess depression in dementia caregivers and has been shown to be sensitive to changes in caregiver depression post intervention. Scores for each item range from 0 (rarely or none of the time) to 3 (most or all of the time), with some items reverse coded. Total scores are calculated by summing all responses and range from 0-60. A higher score is indicative of a worse outcome.
Time Frame: Baseline, 4 month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Media Education and Skill-Building Rehabilitation Int | Usual Care
Number analyzed (Participants) | 8 | 5
score on a scale | -3.00 (4.54) | 1.60 (4.83)

3. Primary Outcome: Change From Baseline Perceived Stress Scale (PSS) at 4 Months
Description: The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale also includes a number of direct queries about current levels of experienced stress. We use a 14 item version of the PSS with a minimum score of 0 and a maximum score of 56. Lower values indicate lower perceived stress while higher values indicate higher perceived stress.
Time Frame: Baseline, 4 month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Media Education and Skill-Building Rehabilitation Int | Usual Care
Number analyzed (Participants) | 8 | 5
score on a scale | -1.00 (9.34) | 3.40 (4.93)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Mobile Media Education and Skill-Building Rehabilitation Int | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2014-03-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT03417219/SAP_000.pdf
  • Study Protocol (2014-08-21): https://cdn.clinicaltrials.gov/large-docs/19/NCT03417219/Prot_001.pdf